CLINICAL TRIAL: NCT05367921
Title: Clinical Validation of CPM#1 Compression Ratio Measurement on Healthy Volunteers
Brief Title: SWISS_EVIDENCE - Compartment Compressibility Monitoring Using CPM#1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Compremium AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SWISS_EVIDENCE
Record Dates: First submitted 2022-04-25; First posted 2022-05-10 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Compartment Syndromes
MeSH Terms: conditions — Compartment Syndromes

STUDY DESIGN:
Masking Description: Investigators will be blinded to the measurement results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPM#1 (Experimental): Compartment compressibility ratio measurement using the CPM#1 device
  Interventions: Device: Measurement of compartment compressibility

INTERVENTIONS:
Device: Measurement of compartment compressibility — Application of the CPM#1 device for compartment compressibility ratio measurement - 4 measurements on both legs of each healthy volunteer will be performed

SUMMARY:
Compartment syndrome is a very serious musculoskeletal disorder, which can lead to potentially devastating consequences, such as limb amputation and life-threatening conditions. It is a well described medical condition considered to be an orthopaedic emergency affecting all ages.

Even though compartment syndrome is a well described medical condition, the appropriate treatment (i.e., fasciotomy to release tissue pressure) is invasive and involves its own risks. Furthermore, and of most critical importance is the timing for the intervention of a fasciotomy. The concerned limb may already have had severe, sometimes even irreversible, tissue damage due to high intra-compartmental pressure within 6 to 10 hours.

The standard diagnostic method for compartment syndrome is an invasive intra-compartmental pressure measurement via insertion of a pressure monitoring device into the muscle compartment. Commercially available intra compartmental pressure monitors have a highly variable intra-observer reproducibility and user errors are common.

Compared to the invasive modalities, the Compremium Compartmental Compressibility Monitoring System (CPM#1) shows promising advantages for the clinical application. Not only is the technology used for the CPM#1 device safe and non-invasive for the patient with minimal training required for the healthcare professionals, but it has also demonstrated high intra- and inter-observer reproducibility (as per bench tests and clinical settings with prototypes, to be confirmed in clinical studies like this one). The use of the CPM#1 device therefore facilitates the measurements, as it is based on pre-existing ultrasound methods and avoids any further risks to the patients compared to invasive compartmental pressure diagnosis methods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Male and female
* Age between 18 and 84

Exclusion Criteria:

* Previous surgery to or fracture of the lower leg
* Peripheral arterial or venous disease
* History of compartment syndrome
* Limb anomalies
* General muscle disorder
* Participants under the influence of excessive alcohol, consumption of narcotics or benzodiazepines prior to procedure
* Participants under the effect of analgesic (< 12 hours)

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Inter-operator reproducibility with 3 raters | During the procedure which should last about 10 min/patient
  Inter-operator reproducibility will be assessed using intra-class correlation coefficients (two-way random effects, single rater, absolute agreement). Three independent raters will conduct one measurement on each of both legs of 21 volunteers.

SECONDARY OUTCOMES:
Intra-operator reproducibility | During the procedure which should last about 10 min/patient
  Intra-operator reproducibility will be assessed using intra-class correlation coefficients (two-way mixed effects, single measurement, absolute agreement). One of the three independent raters will conduct two measurements on 42 legs (21 volunteers).
Participant's reported pain: baseline | Before (5 min before procedure).
  Participant's reported pain will be assessed using a 0-100mm Visual Analogue Scale (VAS) at specific time points.
Participant's reported pain: at highest externally applied pressure | During the procedure (the procedure will last about 10 min/patient)
  Participant's reported pain will be assessed using a 0-100mm Visual Analogue Scale (VAS) at specific time points.
Participant's reported pain: after the procedure | Immediately after procedure (no follow up is planned)
  Participant's reported pain will be assessed using a 0-100mm Visual Analogue Scale (VAS) at specific time points.

OTHER OUTCOMES:
Assessment of adverse events | During the procedure which should last about 10 min/patient
  Safety of the procedure will be assessed by documenting adverse events (description of the adverse events, number of participants).
Assessment of device deficiencies | During the procedure which should last about 10 min/patient
  Safety of the procedure will be assessed by documenting device deficiencies (description)
New risk identification | Within 12 hours after procedure (no follow up is planned)
  Practitioner will be asked to identify risk due to the application of the device in patient care.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Anwander, Dr. med., Principal Investigator — Department für Orthopädie und Traumatologie, Inselspital Bern
Locations (1):
- Universitätsklinik für Orthopädische Chirurgie und Traumatologie Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No